CLINICAL TRIAL: NCT01675882
Title: A Double-blind, Placebo-controlled, Randomized Trial to Study the Viaskin Peanut's Efficacy and Safety for Treating Peanut Allergy in Children and Adults.
Brief Title: Efficacy and Safety of Several Doses of Viaskin Peanut in Adults and Children With Peanut Allergy
Acronym: VIPES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIPES; 2011-002550-32 (EudraCT Number)
Record Dates: First submitted 2012-08-17; First posted 2012-08-30 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Peanut Allergy
Keywords: Food allergy; Immediate hypersensitivity; Whole peanut extract; Allergenic product; Specific Immunotherapy; Epicutaneous Immunotherapy (EPIT)
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Viaskin Peanut 50 mcg (Experimental)
  Interventions: Biological: Viaskin Peanut 50 mcg
- Viaskin Peanut 100 mcg (Experimental)
  Interventions: Biological: Viaskin Peanut 100 mcg
- Viaskin Peanut 250 mcg (Experimental)
  Interventions: Biological: Viaskin Peanut 250 mcg
- Viaskin Placebo (Placebo Comparator)
  Interventions: Biological: Viaskin Placebo

INTERVENTIONS:
Biological: Viaskin Peanut 50 mcg — Subjects epicutaneously administered for 24 hours every 24 hours with a patch containing 50 mcg peanut proteins as whole peanut extract
  Arms: Viaskin Peanut 50 mcg
Biological: Viaskin Peanut 100 mcg — Subjects epicutaneously administered for 24 hours every 24 hours with a patch containing 100 mcg peanut proteins as whole peanut extract
  Arms: Viaskin Peanut 100 mcg
Biological: Viaskin Peanut 250 mcg — Subjects epicutaneously administered for 24 hours every 24 hours with a patch containing 250 mcg peanut proteins as whole peanut extract
  Arms: Viaskin Peanut 250 mcg
Biological: Viaskin Placebo — Subjects epicutaneously administered for 24 hours every 24 hours with a patch containing a matching placebo formulation
  Arms: Viaskin Placebo

SUMMARY:
The objectives of this dose-finding study for the treatment of peanut allergy are:

* To determine the efficacy of 3 doses of Viaskin Peanut (50 mcg ,100 mcg and 250 mcg peanut protein per patch) to significantly desensitize peanut-allergic subjects to peanut after 12 months of treatment.
* To evaluate the safety of a long-term treatment with Viaskin Peanut.

DETAILED DESCRIPTION:
Peanut allergy is a common allergy in the United States, with a prevalence in the general population as high as 1%. Peanut allergy management is based on strict peanut avoidance and injectable epinephrine after the allergic systemic reactions have started. Specific Immunotherapy methods currently available have shown some limitations in their use because of safety issues. Hence, there is an important unmet medical need for efficient and safe treatment of peanut allergy.

DBV Technologies has developed an epicutaneous delivery system, called Viaskin, a method based on delivering precise quantity of the allergen on the upper layers of the skin. Avoiding contact between the allergen and the bloodstream should confer to epicutaneous immunotherapy (EPIT) a higher level of safety as systemic reactions should be circumvented

The VIPES study is a 12-month double-blind, placebo-controlled,randomized trial to study the efficacy and safety of Viaskin Peanut in subjects from 6 to 55 years old with a history of immediate hypersensitive reaction to peanut protein.

The trial will be conducted at sites with investigators and staff trained and experienced in the diagnosis and the management of peanut allergy and anaphylaxis, and who are capable of performing a double-blind placebo-controlled food challenge (DBPCFC) in adult and/or pediatric subjects. Three doses of peanut proteins, i.e. 50 mcg, 100 mcg and 250 mcg will be evaluated for the study. Following the confirmation of peanut allergy at screening, subjects will be randomized in a 1:1:1:1 ratio into four different treatment groups, including 50 mcg, 100 mcg and 250 mcg peanut protein or placebo. Treatment will be comprised of daily applications of Viaskin Peanut or placebo patch for 12 months. Each subject will undergo two DBPCFCs: one at screening and one at Month 12. A follow up visit will be performed 2 weeks after completion of treatment and the last DBPCFC.

ELIGIBILITY:
Inclusion Criteria:

* Peanut-allergic subjects between 6 and 55 years of age, with a well-documented medical history of systemic reactions after ingestion of peanut and currently following a strict peanut-free diet.
* Peanut-specific immunoglobulin E (IgE) level (Phadia CAP-system) > 0.7 kU/L and a positive skin prick test to peanut with a largest wheal diameter ≥ 8 mm
* Positive double-blind placebo-controlled food challenge (DBPCFC) at ≤ 300 mg of peanut proteins: the eliciting dose of peanut proteins during the DBPCFC is capped at 300 mg, i.e. subjects must react to peanut before reaching or at the dose of 300 mg peanut proteins.
* Negative pregnancy test for women of childbearing potential. Females of childbearing age must use effective methods of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the study. Sexual abstinence will be accepted as an effective method of contraception for girls below 15 years of age.
* Ability to perform spirometry maneuvers in accordance with the American Thoracic Society guidelines (2005) for subjects 9 years of age and above Subjects below 9 years of age can perform peak expiratory flow (PEF) instead.
* Willing to comply with all study requirements during their participation in the study.
* Provide signed informed consent and assent as appropriate.

Exclusion Criteria:

* Subjects with a history of severe anaphylaxis to peanut with the following symptoms: hypotension, hypoxia, neurological compromise (collapse, loss of consciousness or incontinence).
* Pregnancy or lactation.
* FEV1 <80% of the predicted value at screening for subjects 9 years of age and above. PEF < 80% of predicted for subjects below 9 years of age.
* Subjects who did not react at or below the dose of 300 mg of peanut proteins during the DBPCFC at screening.
* Known allergy or known hypersensitivity to placebo excipients either of the Viaskin patches or of the food challenge formulas.
* Subjects reacting objectively to the placebo formula at screening.
* Severe reaction during the screening food challenge, defined as need for intubation, hypotension persisting after epinephrine administration, or the need for more than two doses of epinephrine.
* Inability to discontinue short-acting antihistamines for three days or long-acting antihistamines for five to seven days (depending on half-life) prior to skin prick testing or food challenges.
* Subjects treated with systemic long-acting corticosteroids (depot corticosteroids) within 12 weeks prior to the screening visit and/or systemic short-acting corticosteroid within 4 weeks prior to the screening visit or any systemic corticosteroid at screening.
* Subjects with asthma defined as follows:

  1. uncontrolled persistent asthma by National Asthma Education and Prevention Program Asthma guidelines (2007) or by Global Initiative for Asthma (2011) or being treated with combination therapy of medium dose inhaled corticosteroid with a long acting inhaled β2-agonists;
  2. at least two systemic corticosteroid courses for asthma in the past year or one oral corticosteroid course for asthma in the past three months;
  3. prior intubation for asthma in the past two years.
* Subjects on β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, calcium channel blockers or tricyclic antidepressant therapy.
* Subjects undergoing any type of immunotherapy to any food within one year prior to the screening visit.
* Subjects presently on aeroallergen immunotherapy and unwilling or unable to discontinue.
* Subjects currently treated with anti-tumor necrosis factor drugs or anti-IgE drugs (such as omalizumab) or any biologic immunomodulatory therapy within one year prior to the screening visit.
* Allergy or known history of reaction to Tegaderm®.
* Subjects suffering from generalized dermatologic diseases (e.g. severe atopic dermatitis, uncontrolled generalized eczema, keratosis pilaris, ichthyosis vulgaris) with no intact skin zones to apply the patches.
* Any disorder in which epinephrine is contraindicated such as coronary artery disease, uncontrolled hypertension, or serious ventricular arrhythmias.
* Participation in another clinical intervention study in the three months prior to the screening visit.
* Subjects on any experimental drugs or treatments.

Other inclusion/exclusion criteria may apply.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (10):
  - University of California, Rady Childrens Hospital, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens' Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - ASTHMA, Inc., Seattle, Washington
- Canada (4):
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Asthma Research Institute, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario
  - Centre de Recherche Appliquée en Asthme et Allergie de Québec, Sainte-Foy, Quebec
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux, Hôpital Pellegrin, Bordeaux
  - Hôpital Saint Vincent de Paul, Lille
  - GCS des hôpitaux pédiatriques, Nice
  - Hôpital Necker, Paris
  - Nouvel Hôpital Civil, Strasbourg
  - Hôpitaux De Brabois, Vandœuvre-lès-Nancy
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (2):
  - Szpital Uniwersytecki nr2, Bydgoszcz
  - Szpital Kliniczny UM, Lodz

REFERENCES:
- [Derived] Lewis MO, Brown-Whitehorn TF, Cianferoni A, Rooney C, Spergel JM. Peanut-allergic patient experiences after epicutaneous immunotherapy: peanut consumption and impact on QoL. Ann Allergy Asthma Immunol. 2019 Jul;123(1):101-103. doi: 10.1016/j.anai.2019.04.006. Epub 2019 Apr 10. No abstract available. PMID 30978404
- [Derived] Sampson HA, Shreffler WG, Yang WH, Sussman GL, Brown-Whitehorn TF, Nadeau KC, Cheema AS, Leonard SA, Pongracic JA, Sauvage-Delebarre C, Assa'ad AH, de Blay F, Bird JA, Tilles SA, Boralevi F, Bourrier T, Hebert J, Green TD, Gerth van Wijk R, Knulst AC, Kanny G, Schneider LC, Kowalski ML, Dupont C. Effect of Varying Doses of Epicutaneous Immunotherapy vs Placebo on Reaction to Peanut Protein Exposure Among Patients With Peanut Sensitivity: A Randomized Clinical Trial. JAMA. 2017 Nov 14;318(18):1798-1809. doi: 10.1001/jama.2017.16591. PMID 29136445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase IIb, placebo-controlled study was conducted in participants aged 6 to 55 years old with peanut allergy at 22 study centers in 5 countries (Canada, France, Netherlands, Poland and USA) between 31 July 2012 and 31 July 2014. All participants who completed the VIPES study up to Visit 11 (inclusive) were eligible for participation in the follow-up study (OLFUS-VIPES).
Pre-assignment Details: Study had a 4-week screening period, 52-week treatment period and 2-week follow-up period. A total of 221 participants were randomized in a 1:1:1:1 ratio into 4 treatment groups (50 micrograms [μg], 100 μg, 250 μg peanut proteins and placebo). Each participant underwent dose-escalating double-blind, placebo-controlled food challenge (DBPCFC) at screening and Month 12. At screening, a dose-escalating DBPCFC confirmed peanut allergy to an eliciting dose <=300 milligrams (mg) peanut protein.
Groups:
- Viaskin Peanut 50 μg: Participants applied 1 new Viaskin® Peanut (DBV712) 50 μg patch on intact skin for 24 hours daily for 12 months. To better ensure the safety of the patch at the initiation of treatment, the application duration was progressively increased to a duration of 24 hours daily over a 21-day graduated dosing period.
- Viaskin Peanut 100 μg: Participants applied 1 new Viaskin Peanut 100 μg patch on intact skin for 24 hours daily for 12 months. To better ensure the safety of the patch at the initiation of treatment, the application duration was progressively increased to a duration of 24 hours daily over a 21-day graduated dosing period.
- Viaskin Peanut 250 μg: Participants applied 1 new Viaskin Peanut 250 μg patch on intact skin for 24 hours daily for 12 months. To better ensure the safety of the patch at the initiation of treatment, the application duration was progressively increased to a duration of 24 hours daily over a 21-day graduated dosing period.
- Placebo: Participants applied 1 new placebo patch on intact skin for 24 hours daily for 12 months. To better ensure the safety of the patch at the initiation of treatment, the application duration was progressively increased to a duration of 24 hours daily over a 21-day graduated dosing period.
Period: Overall Study
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Started | 53 | 56 | 56 | 56
Completed | 51 | 49 | 53 | 54
Not Completed | 2 | 7 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Participant unwilling to continue | 2 | 4 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Viaskin Peanut 50 μg: Participants applied 1 new Viaskin Peanut 50 μg patch on intact skin for 24 hours daily for 12 months. To better ensure the safety of the patch at the initiation of treatment, the application duration was progressively increased to a duration of 24 hours daily over a 21-day graduated dosing period.
- Total: Total of all reporting groups
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo | Total
Number analyzed (Participants) | 53 | 56 | 56 | 56 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.3 (6.72) | 13.9 (6.66) | 13.6 (7.48) | 12.5 (6.84) | 13.1 (6.92)
Age, Customized [Count of Participants; unit: Participants]
  Children (6-11 years) | 28 | 26 | 28 | 31 | 113
  Adolescents (12-17 years) | 18 | 19 | 18 | 18 | 73
  Adults (18-55 years) | 7 | 11 | 10 | 7 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 18 | 20 | 83
  Male | 31 | 33 | 38 | 36 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The ethnicity of the participants at French local sites was not collected as it was not applicable as per local law. As such, these participants are included in the category of 'Not applicable'.
  Participants
    Caucasian | 39 | 33 | 32 | 31 | 135
    Black | 1 | 2 | 0 | 2 | 5
    Hispanic | 1 | 0 | 0 | 2 | 3
    Asian | 3 | 9 | 10 | 5 | 27
    Other | 2 | 4 | 4 | 4 | 14
    Not applicable | 7 | 8 | 10 | 12 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 16 | 19 | 19 | 17 | 71
  Netherlands | 2 | 3 | 2 | 2 | 9
  United States | 28 | 26 | 24 | 25 | 103
  Poland | 0 | 0 | 1 | 0 | 1
  France | 7 | 8 | 10 | 12 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders at Month 12; Analyzed in Overall Population
Description: A treatment responder was defined as a participant with a peanut protein eliciting dose equal to or greater than 1,000 mg peanut proteins based on the results of the DBPCFC after 12 months of treatment or a participant with a >=10-fold increase of the eliciting dose at 12 months, compared to the initial eliciting dose. For participants with missing treatment response at Month 12, last observation carried forward (LOCF) imputation was used (i.e., participants were considered as non-responders).
Time Frame: At Month 12
Population: The full analysis set included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
percentage of participants | 45.3 [31.56 to 59.55] | 41.1 [28.10 to 55.02] | 50.0 [36.34 to 63.66] | 25.0 [14.39 to 38.37]
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; The three pair-wise comparisons of viaskin peanut versus placebo were analyzed using the Bonferroni stepwise procedure, keeping the overall false-positive (alpha) risk below 5%. The comparison of viaskin peanut 250 µg versus placebo is statistically significant at p<0.05. The subsequent comparison of viaskin peanut 100 µg versus placebo is not statistically significant at p<0.05. Thus, no conclusion can be made on the comparison of viaskin peanut 50 µg vs placebo; Test type: Superiority; p = 0.0292, Fisher Exact; Relative risk = 1.81, 95% CI 2-sided [1.05 to 3.11]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; The three pair-wise comparisons of viaskin peanut versus placebo were analyzed using the Bonferroni stepwise procedure, keeping the overall false-positive (alpha) risk below 5%. The comparison of viaskin peanut 250 µg versus placebo is statistically significant at p<0.05. The subsequent comparison of viaskin peanut 100 µg versus placebo is not statistically significant at p<0.05; Test type: Superiority; p = 0.1074, Fisher Exact; Relative risk = 1.64, 95% CI 2-sided [0.95 to 2.85]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; The three pair-wise comparisons of viaskin peanut versus placebo were analyzed using the Bonferroni stepwise procedure, keeping the overall false-positive (alpha) risk below 5%. The comparison of viaskin peanut 250 µg versus placebo is statistically significant at p<0.05; Test type: Superiority; p = 0.0108, Fisher Exact; Relative risk = 2.00, 95% CI 2-sided [1.18 to 3.38]

2. Secondary Outcome: Percentage of Treatment Responders at Month 12; Analyzed in Children (6-11 Years of Age)
Description: A treatment responder was defined as a participant with a peanut protein eliciting dose equal to or greater than 1,000 mg peanut proteins based on the results of the DBPCFC after 12 months of treatment or a participant with a >=10-fold increase of the eliciting dose at 12 months, compared to the initial eliciting dose. For participants with missing treatment response at Month 12, LOCF imputation was used (i.e., participants were considered as non-responders).
Time Frame: At Month 12
Population: The full analysis set included all participants who were randomized. Only participants in the range of 6-11 years of age are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 28 | 26 | 28 | 31
percentage of participants | 57.1 [37.18 to 75.54] | 46.2 [26.59 to 66.63] | 53.6 [33.87 to 72.49] | 19.4 [7.45 to 37.47]
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; Test type: Superiority; p = 0.0035, Fisher Exact; Relative risk = 2.95, 95% CI 2-sided [1.34 to 6.49]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; Test type: Superiority; p = 0.0453, Fisher Exact; Relative risk = 2.38, 95% CI 2-sided [1.04 to 5.47]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; Test type: Superiority; p = 0.0076, Fisher Exact; Relative risk = 2.77, 95% CI 2-sided [1.25 to 6.14]

3. Secondary Outcome: Percentage of Treatment Responders at Month 12; Analyzed in Adolescents (12-17 Years of Age)
Description: as for outcome 2
Time Frame: At Month 12
Population: The full analysis set included all participants who were randomized. Only participants in the range of 12-17 years of age are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 18 | 19 | 18 | 18
percentage of participants | 33.3 [13.34 to 59.01] | 10.5 [1.30 to 33.14] | 38.9 [17.30 to 64.25] | 22.2 [6.41 to 47.64]
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; Test type: Superiority; p = 0.7112, Fisher Exact; Relative risk = 1.50, 95% CI 2-sided [0.51 to 4.43]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; Test type: Superiority; p = 0.4048, Fisher Exact; Relative risk = 0.47, 95% CI 2-sided [0.10 to 2.28]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; Test type: Superiority; p = 0.4705, Fisher Exact; Relative risk = 1.75, 95% CI 2-sided [0.62 to 4.95]

4. Secondary Outcome: Percentage of Treatment Responders at Month 12; Analyzed in Adults (18-55 Years of Age)
Description: as for outcome 2
Time Frame: At Month 12
Population: The full analysis set included all participants who were randomized. Only participants in the range of 18-55 years of age are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 7 | 11 | 10 | 7
percentage of participants | 28.6 [3.67 to 70.96] | 81.8 [48.22 to 97.72] | 60.0 [26.24 to 87.84] | 57.1 [18.41 to 90.10]
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; Test type: Superiority; p = 0.5921, Fisher Exact; Relative risk = 0.50, 95% CI 2-sided [0.13 to 1.90]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; Test type: Superiority; p = 0.3260, Fisher Exact; Relative risk = 1.43, 95% CI 2-sided [0.71 to 2.88]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; Test type: Superiority; p = 1.0000, Fisher Exact; Relative risk = 1.05, 95% CI 2-sided [0.46 to 2.38]

5. Secondary Outcome: Mean Eliciting Doses of Peanut Proteins at Month 12; Analyzed in Overall Population
Description: The peanut protein eliciting dose was defined as the first dose of peanut protein administered to the participant during the DBPCFC procedure which caused an objective allergic reaction. This was capped to 300 mg at the screening DBPCFC and to 2000 mg at the Month 12 DBPCFC. For participants with missing treatment response at Month 12, LOCF imputation was used (i.e., participants were considered as non-responders).
Time Frame: At Month 12
Population: The full analysis set included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
mg | 453.8 (608.16) | 539.7 (659.31) | 621.4 (715.03) | 283.7 (482.04)
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; The least squares (LS) mean for any given treatment group is the estimated mean peanut protein eliciting dose for a participant in that treatment group with the mean value for all baseline covariates in the analysis set; Test type: Superiority; p = 0.0607, ANCOVA — P-value was based on type III sum of squares from analysis of covariance (ANCOVA) model on log transformed values for peanut protein eliciting dose at Month 12, including treatment group, baseline eliciting dose, age-strata and country as covariates; Difference in LS mean = 70.2, 95% CI 2-sided [-2.41 to 193.69]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; The LS mean for any given treatment group is the estimated mean peanut protein eliciting dose for a participant in that treatment group with the mean value for all baseline covariates in the analysis set; Test type: Superiority; p = 0.0150, ANCOVA — P-value was based on type III sum of squares from an ANCOVA model on log transformed values for the peanut protein eliciting dose at Month 12, including treatment group, baseline eliciting dose, age-strata and country as covariates; Difference in LS mean = 97.5, 95% CI 2-sided [14.45 to 237.82]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 242.2, 95% CI 2-sided [100.03 to 482.65]

6. Secondary Outcome: Mean Eliciting Doses of Peanut Proteins at Month 12; Analyzed in Children (6-11 Years of Age)
Description: The peanut protein eliciting dose was defined as the first dose of peanut protein administered to the participant during the DBPCFC procedure which caused an objective allergic reaction. This was capped to 300 mg at screening DBPCFC and to 2000 mg at the Month 12 DBPCFC. For participants with missing treatment response at Month 12, LOCF imputation was used (i.e., participants were considered as non-responders).
Time Frame: At Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 28 | 26 | 28 | 31
mg | 397.1 (510.13) | 441.2 (511.26) | 652.5 (766.93) | 160.5 (244.00)
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0372, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 73.9, 95% CI 2-sided [2.96 to 225.85]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0143, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 96.7, 95% CI 2-sided [12.92 to 278.11]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 260.3, 95% CI 2-sided [89.83 to 625.95]

7. Secondary Outcome: Mean Eliciting Doses of Peanut Proteins at Month 12; Analyzed in Adolescents (12-17 Years of Age)
Description: as for outcome 6
Time Frame: At Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 18 | 19 | 18 | 18
mg | 501.7 (726.14) | 281.6 (472.47) | 573.9 (716.01) | 331.8 (511.62)
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.6596, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 26.1, 95% CI 2-sided [-59.58 to 236.00]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.8702, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 8.9, 95% CI 2-sided [-65.90 to 189.96]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.0630, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 158.9, 95% CI 2-sided [-5.50 to 562.31]

8. Secondary Outcome: Mean Eliciting Doses of Peanut Proteins at Month 12; Analyzed in Adults (18-55 Years of Age)
Description: as for outcome 6
Time Frame: At Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 7 | 11 | 10 | 7
mg | 557.1 (711.47) | 1218.5 (822.74) | 620.0 (619.68) | 705.7 (893.01)
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.6776, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = -80.2, 95% CI 2-sided [-237.22 to 782.24]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.5068, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 158.8, 95% CI 2-sided [-166.10 to 1478.83]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.7972, ANCOVA — [p-value comment as in outcome 5, analysis 2]; Difference in LS mean = 53.8, 95% CI 2-sided [-193.90 to 1085.38]

9. Secondary Outcome: Mean Cumulative Reactive Dose of Peanut Proteins at Month 12; Analyzed in Overall Population
Description: The peanut protein cumulative reactive dose was defined as the sum of all peanut protein doses up to and including the eliciting dose ingested during the peanut challenge. For participants with missing treatment response at Month 12, LOCF imputation was used (i.e., participants were considered as non-responders).
Time Frame: At Month 12
Population: The full analysis set included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
mg | 730.8 (1020.53) | 863.5 (1120.43) | 1010.6 (1223.85) | 451.4 (807.13)
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; The LS mean for any given treatment group was the estimated mean peanut protein cumulative reactive dose for a participant in that treatment group with the mean value for all baseline covariates in the analysis set; Test type: Superiority; p = 0.0444, ANCOVA — P-value was based on type III sum of squares from an ANCOVA model on log transformed values for cumulative reactive dose at Month 12, including treatment group, baseline cumulative reactive dose, age-strata and country as covariates; Difference in LS mean = 120.0, 95% CI 2-sided [2.30 to 321.80]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0175, ANCOVA — P-value was based on type III sum of squares from an ANCOVA model on log transformed values for the cumulative reactive dose at Month 12, including treatment group, baseline cumulative reactive dose, age-strata and country as covariates; Difference in LS mean = 147.6, 95% CI 2-sided [19.67 to 365.51]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 9, analysis 2]; Difference in LS mean = 386.0, 95% CI 2-sided [159.67 to 771.16]

10. Secondary Outcome: Change From Baseline in Severity of Symptoms Based on the Oral Food Challenge (OFC) Symptom Score Sheet at Month 12; Analyzed in Overall Population
Description: The symptoms of erythematous rash, pruritus, urticaria/angioedema, rash, sneezing/itching, nasal congestion, rhinorrhea, laryngeal symptoms (example, throat clearing, occasional cough, hoarseness, frequent dry cough, inspiratory stridor), wheezing, subjective complaints, objective complaints and cardiovascular symptoms (example, color change, weakness, dizziness, mental status change, tachycardia, decreased blood pressure, etc) were observed. The OFC score ranges from 0 to 3 for each symptom (0=Absent, 1=mild, 2=moderate or 3=severe). The total symptom score for each participant was calculated. Higher scores indicate worst outcome. For participants with missing treatment response at Month 12, LOCF imputation was used (i.e., participants were considered as non-responders).
Time Frame: Baseline and Month 12
Population: The full analysis set included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
units on a scale | -1.9 (4.79) | -0.9 (4.21) | 0.2 (4.65) | -1.4 (4.35)
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; The LS mean for any given treatment group is the estimated mean OFC score for a participant in that treatment group with the mean value for all baseline covariates in the analysis set; Test type: Superiority; p = 0.2510, ANCOVA — P-value was based on type III sum of squares from an ANCOVA model on log transformed values for the OFC symptom scores at Month 12, including treatment group, Baseline OFC symptom scores, age-strata and country as covariates; Difference in LS mean = -0.6, 95% CI 2-sided [-1.55 to 0.52]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.6820, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Difference in LS mean = -0.2, 95% CI 2-sided [-1.24 to 1.05]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.2117, ANCOVA — [p-value comment as in outcome 10, analysis 1]; Difference in LS mean = 0.8, 95% CI 2-sided [-0.42 to 2.47]

11. Secondary Outcome: Number of Participants With an Average Wheal Diameter Ratio ≤0.5 and >0.5 at Each Skin Prick Test Dilution at Months 3, 6 and 12; Analyzed in Overall Population
Description: The mean wheal diameter of skin prick test (sum of the orthogonal diameters divided by 2) at each time point is calculated for the 5 skin prick tests at baseline and at each time point, i.e., Months 3, 6 and 12: undiluted, diluted 1:10 millimeter (mm), diluted 1:100 (mm), diluted 1:1,000 (mm), diluted 1:10,000 (mm). The ratio of the mean wheal diameter at each time point for a specific dilution versus the baseline value for that specific dilution was calculated and classified as <=0.5 or >0.5, allowing to assess the number of participants of those mean wheal diameters that have been at least halved from the baseline value.
Time Frame: Baseline and Months 3, 6 and 12
Population: The full analysis set included all participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
Participants
  Month 3: undiluted; <= 0.5 | 7 | 9 | 5 | 4
  Month 3: undiluted; > 0.5 | 46 | 47 | 51 | 52
  Month 3: diluted (1:10); <= 0.5 | 10 | 5 | 8 | 4
  Month 3: diluted (1:10); > 0.5 | 43 | 51 | 48 | 52
  Month 3: diluted (1:100); <= 0.5 | 13 | 12 | 15 | 6
  Month 3: diluted (1:100); > 0.5 | 39 | 43 | 41 | 50
  Month 3: diluted (1:1000); <= 0.5 | 13 | 15 | 24 | 12
  Month 3: diluted (1:1000); > 0.5 | 35 | 35 | 28 | 40
  Month 3: diluted (1:10000); <= 0.5 | 21 | 17 | 22 | 15
  Month 3: diluted (1:10000); > 0.5 | 21 | 18 | 20 | 24
  Month 6: undiluted; <= 0.5 | 14 | 7 | 7 | 2
  Month 6: undiluted; > 0.5 | 39 | 49 | 49 | 54
  Month 6: diluted (1:10); <= 0.5 | 9 | 10 | 9 | 5
  Month 6: diluted (1:10); > 0.5 | 44 | 46 | 47 | 51
  Month 6: diluted (1:100); <= 0.5 | 15 | 16 | 14 | 4
  Month 6: diluted (1:100); > 0.5 | 37 | 39 | 42 | 52
  Month 6: diluted (1:1000); <= 0.5 | 15 | 11 | 23 | 11
  Month 6: diluted (1:1000); > 0.5 | 33 | 39 | 29 | 41
  Month 6: diluted (1:10000); <= 0.5 | 21 | 15 | 22 | 14
  Month 6: diluted (1:10000); > 0.5 | 21 | 20 | 20 | 25
  Month 12: undiluted; <= 0.5 | 8 | 4 | 7 | 2
  Month 12: undiluted; > 0.5 | 45 | 52 | 49 | 54
  Month 12: diluted (1:10); <= 0.5 | 10 | 6 | 15 | 3
  Month 12: diluted (1:10); > 0.5 | 43 | 50 | 41 | 53
  Month 12: diluted (1:100); <= 0.5 | 11 | 14 | 13 | 7
  Month 12: diluted (1:100); > 0.5 | 41 | 41 | 43 | 49
  Month 12: diluted (1:1000); <= 0.5 | 14 | 9 | 18 | 8
  Month 12: diluted (1:1000); > 0.5 | 34 | 41 | 34 | 44
  Month 12: diluted (1:10000); <= 0.5 | 22 | 14 | 24 | 13
  Month 12: diluted (1:10000); > 0.5 | 20 | 21 | 18 | 26

12. Secondary Outcome: Change From Baseline in Peanut-Specific Immunoglobulin E (IgE) at Months 3, 6 and 12; Analyzed in Overall Population
Description: Venous blood samples were taken for assessment of the peanut-specific IgE at 3, 6 and 12 months. Results are presented using multiple imputation to replace missing values.
Time Frame: Baseline and Months 3, 6 and 12
Population: The full analysis set included all participants who were randomized.
Measure: Median (Full Range); unit: kilo units per liter (kU/L)
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
kilo units per liter (kU/L)
  Month 3 | 32.3 [-375 to 676] | 29.9 [-118 to 1243] | 50.7 [-91 to 794] | 2.8 [-117 to 445]
  Month 6 | 8.8 [-158 to 348] | 22.0 [-65 to 1464] | 29.5 [-93 to 747] | -1.1 [-363 to 79]
  Month 12 | -0.2 [-211 to 305] | 4.9 [-146 to 245] | 5.2 [-382 to 598] | -1.4 [-327 to 93]
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; The LS mean for any given treatment group was the estimated mean for a participant in that treatment group with the mean value for all Baseline covariates in the analysis set; Test type: Superiority; p = 0.0337, ANCOVA — P-value was based on type III sum of squares from an ANCOVA model on log transformed values for the immunological marker at Month 12, including treatment group, Baseline marker, age-strata and country as covariates; Difference in LS mean = 17.4, 95% CI 2-sided [1.17 to 38.82]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0020, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Difference in LS mean = 26.2, 95% CI 2-sided [8.38 to 49.45]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0120, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Difference in LS mean = 20.0, 95% CI 2-sided [3.85 to 40.91]

13. Secondary Outcome: Change From Baseline in Peanut-Specific IgE at Months 3, 6 and 12; Analyzed in Children (6-11 Years of Age)
Description: as for outcome 12
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 2
Measure: Median (Full Range); unit: kU/L
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 28 | 26 | 28 | 31
kU/L
  Month 3 | 63.6 [-375 to 676] | 63.1 [-27 to 1243] | 50.7 [-16 to 794] | 4.1 [-117 to 445]
  Month 6 | 10.6 [-55 to 348] | 48.7 [-9 to 1464] | 21.2 [-70 to 291] | -1.8 [-363 to 79]
  Month 12 | -3.1 [-211 to 305] | 3.5 [-146 to 150] | 1.0 [-136 to 485] | -12.0 [-327 to 59]

14. Secondary Outcome: Change From Baseline in Peanut-Specific IgE at Months 3, 6 and 12; Analyzed in Adolescents (12-17 Years of Age)
Description: as for outcome 12
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: kU/L
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 18 | 19 | 18 | 18
kU/L
  Month 3 | 11.5 [-99 to 248] | 62.0 [-118 to 303] | 135.5 [0 to 552] | 4.8 [-17 to 232]
  Month 6 | 6.0 [-158 to 170] | 24.2 [-65 to 239] | 90.0 [-10 to 440] | 0.0 [-43 to 75]
  Month 12 | 5.2 [-49 to 199] | 24.9 [-98 to 163] | 39.4 [-382 to 434] | 1.0 [-31 to 93]

15. Secondary Outcome: Change From Baseline in Peanut-Specific IgE at Months 3, 6 and 12; Analyzed in Adults (18-55 Years of Age)
Description: as for outcome 12
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 4
Measure: Median (Full Range); unit: kU/L
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 7 | 11 | 10 | 7
kU/L
  Month 3 | 65.3 [-76 to 183] | 12.3 [-1 to 169] | 3.1 [-91 to 471] | 0.1 [-34 to 13]
  Month 6 | 34.4 [-0 to 214] | 3.6 [-4 to 377] | 1.6 [-93 to 747] | -0.2 [-42 to 40]
  Month 12 | 22.3 [-25 to 163] | 0.3 [-9 to 245] | -2.0 [-148 to 598] | 0.9 [-107 to 39]

16. Secondary Outcome: Change From Baseline in Peanut-Specific Immunoglobulin G Subtype 4 (IgG4) at Months 3, 6 and 12; Analyzed in Overall Population
Description: Venous blood samples were taken for assessment of the peanut-specific IgG4 at 3, 6 and 12 months. Results are presented using multiple imputation to replace missing values.
Time Frame: Baseline and Months 3, 6 and 12
Population: The full analysis set included all participants who were randomized.
Measure: Median (Full Range); unit: mg per liter (mg/L)
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 53 | 56 | 56 | 56
mg per liter (mg/L)
  Month 3 | 0.4 [-1 to 6] | 0.4 [-18 to 4] | 0.8 [-1 to 14] | 0.0 [-3 to 2]
  Month 6 | 0.8 [-2 to 6] | 0.8 [-19 to 8] | 1.4 [-6 to 19] | 0.0 [-2 to 3]
  Month 12 | 1.0 [-2 to 12] | 0.9 [-9 to 10] | 1.6 [-3 to 17] | 0.0 [-3 to 1]
Statistical Analysis 1: Comparison: Viaskin Peanut 50 μg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Difference in LS mean = 1.2, 95% CI 2-sided [0.72 to 1.90]
Statistical Analysis 2: Comparison: Viaskin Peanut 100 μg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Difference in LS mean = 1.3, 95% CI 2-sided [0.79 to 2.01]
Statistical Analysis 3: Comparison: Viaskin Peanut 250 μg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; Difference in LS mean = 2.1, 95% CI 2-sided [1.39 to 3.11]

17. Secondary Outcome: Change From Baseline in Peanut-Specific IgG4 at Months 3, 6 and 12; Analyzed in Children (6-11 Years of Age)
Description: as for outcome 16
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/L
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 28 | 26 | 28 | 31
mg/L
  Month 3 | 0.6 [-1 to 6] | 0.4 [-18 to 4] | 1.7 [-1 to 14] | 0.0 [-1 to 1]
  Month 6 | 1.1 [-2 to 6] | 1.1 [-19 to 8] | 4.4 [0 to 19] | -0.1 [-1 to 2]
  Month 12 | 2.0 [-2 to 12] | 1.6 [-9 to 10] | 6.3 [-1 to 17] | -0.0 [-2 to 1]

18. Secondary Outcome: Change From Baseline in Peanut-Specific IgG4 at Months 3, 6 and 12; Analyzed in Adolescents (12-17 Years of Age)
Description: as for outcome 16
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 3
Measure: Median (Full Range); unit: mg/L
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 18 | 19 | 18 | 18
mg/L
  Month 3 | 0.1 [-0 to 2] | 0.6 [-0 to 2] | 0.7 [-0 to 4] | 0.1 [-3 to 2]
  Month 6 | 0.3 [-1 to 3] | 0.8 [0 to 2] | 0.7 [-6 to 6] | 0.1 [-2 to 3]
  Month 12 | 0.4 [-1 to 8] | 0.7 [-1 to 3] | 0.9 [-3 to 9] | 0.1 [-3 to 1]

19. Secondary Outcome: Change From Baseline in Peanut-Specific IgG4 at Months 3, 6 and 12; Analyzed in Adults (18-55 Years of Age)
Description: as for outcome 16
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 4
Measure: Median (Full Range); unit: mg/L
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
Number analyzed (Participants) | 7 | 11 | 10 | 7
mg/L
  Month 3 | 0.2 [0 to 3] | 0.5 [-0 to 2] | 0.4 [-0 to 1] | 0.1 [-0 to 0.4]
  Month 6 | 0.5 [-0 to 3] | 0.5 [-0 to 1] | 0.6 [-0 to 6] | 0.0 [-0 to 1]
  Month 12 | 0.6 [0 to 3] | 0.3 [0 to 1] | 0.9 [-0 to 8] | 0.1 [-0 to 0.4]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Day 1, throughout the 52-week treatment period and additional 2-week follow-up period. Overall time frame of up to 54 weeks.
Description: The safety analysis set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Viaskin Peanut 50 μg | Viaskin Peanut 100 μg | Viaskin Peanut 250 μg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/56 | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/56 | 2/56 | 0/56
Other Adverse Events (participants affected / at risk) | 53/53 | 55/56 | 56/56 | 51/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viaskin Peanut 50 μg (N=53) | Viaskin Peanut 100 μg (N=56) | Viaskin Peanut 250 μg (N=56) | Placebo (N=56)
Anaphylactic reaction (Immune system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viaskin Peanut 50 μg (N=53) | Viaskin Peanut 100 μg (N=56) | Viaskin Peanut 250 μg (N=56) | Placebo (N=56)
Eye swelling (Eye disorders) | 1 (1) | 2 (3) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (9) | 3 (6) | 2 (2) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 7 (8)
Vomiting (Gastrointestinal disorders) | 5 (8) | 3 (3) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (6) | 1 (1) | 3 (3) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (2)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Application site erythema (General disorders) | 39 (53) | 33 (68) | 32 (61) | 14 (21)
Application site pruritus (General disorders) | 18 (23) | 23 (52) | 23 (38) | 7 (15)
Pyrexia (General disorders) | 9 (15) | 7 (8) | 6 (7) | 10 (12)
Application site eczema (General disorders) | 7 (9) | 8 (12) | 10 (17) | 1 (1)
Application site swelling (General disorders) | 5 (6) | 8 (8) | 12 (15) | 3 (5)
Application site papules (General disorders) | 6 (6) | 8 (8) | 9 (12) | 1 (1)
Application site dermatitis (General disorders) | 5 (5) | 6 (6) | 8 (9) | 3 (4)
Application site rash (General disorders) | 7 (11) | 1 (1) | 1 (2) | 6 (6)
Application site reaction (General disorders) | 2 (2) | 2 (4) | 4 (6) | 3 (6)
Application site urticaria (General disorders) | 2 (3) | 5 (6) | 5 (7) | 2 (2)
Application site discolouration (General disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Application site irritation (General disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Application site oedema (General disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Application site pain (General disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Application site dryness (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Food allergy (Immune system disorders) | 8 (11) | 11 (22) | 7 (11) | 10 (14)
Seasonal allergy (Immune system disorders) | 5 (9) | 3 (6) | 6 (7) | 3 (5)
Hypersensitivity (Immune system disorders) | 4 (5) | 3 (3) | 1 (1) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 14 (23) | 11 (18) | 12 (17) | 12 (25)
Nasopharyngitis (Infections and infestations) | 12 (13) | 9 (17) | 10 (15) | 18 (30)
Gastroenteritis (Infections and infestations) | 2 (3) | 3 (4) | 6 (6) | 8 (8)
Ear infection (Infections and infestations) | 3 (5) | 5 (7) | 1 (1) | 5 (6)
Gastroenteritis viral (Infections and infestations) | 6 (8) | 4 (4) | 4 (4) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 3 (4) | 4 (5) | 2 (2) | 3 (4)
Viral infection (Infections and infestations) | 1 (1) | 5 (6) | 1 (1) | 4 (6)
Viral upper respiratory tract infection (Infections and infestations) | 2 (5) | 2 (3) | 1 (2) | 3 (4)
Pharyngitis (Infections and infestations) | 5 (8) | 1 (1) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3) | 2 (3)
Rhinitis (Infections and infestations) | 0 (0) | 3 (5) | 1 (1) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 11 (17) | 8 (16) | 8 (14) | 13 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (7) | 5 (5) | 5 (15)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (14) | 1 (1) | 6 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 5 (7) | 7 (7) | 6 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 8 (9) | 4 (4) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (4) | 7 (7) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (7) | 3 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 2 (2) | 0 (0) | 4 (9)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 8 (16) | 3 (5) | 8 (9) | 8 (18)
Eczema (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 5 (7) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 5 (5) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes